CLINICAL TRIAL: NCT03787186
Title: A Phase 1, Open-label, Single-center Study to Investigate the Pharmacokinetics and Metabolism of GLPG1690 in Healthy Male Subjects Following Single Intravenous GLPG1690 Microtracer and Oral [14C]-GLPG1690 Administrations.
Brief Title: A Study in Healthy Male Volunteers to Look at How the Test Medicine GLPG1690 is Taken up by the Body When Given by Mouth and Into a Vein as an Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG1690-CL-107
Record Dates: First submitted 2018-12-17; First posted 2018-12-26 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG1690 oral and IV (Experimental): GLPG1690 film-coated tablets followed by [14C]-GLPG1690 solution for infusion
  Interventions: Drug: GLPG1690 film-coated tablets; Drug: [14C]-GLPG1690 solution for infusion
- [14C]-GLPG1690 capsules (Experimental): [14C]-GLPG1690 capsules
  Interventions: Drug: [14C]-GLPG1690 capsules

INTERVENTIONS:
Drug: GLPG1690 film-coated tablets — a single oral dose of GLPG1690
  Arms: GLPG1690 oral and IV
Drug: [14C]-GLPG1690 solution for infusion — a 15-minute IV infusion [14C]-GLPG1690
  Arms: GLPG1690 oral and IV
Drug: [14C]-GLPG1690 capsules — single oral dose of [14C]-GLPG1690
  Arms: [14C]-GLPG1690 capsules

SUMMARY:
The sponsor wants to investigate how well the test medicine is taken up by the body when given orally (by mouth) as a tablet or capsule and as a solution for infusion (into a vein). The capsule and the solution will be radiolabelled. 'Radiolabelled' means that the test medicine has a radioactive component which helps us to track where the test medicine is in the body.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with the clinical study protocol (CSP) requirements and sign the informed consent form (ICF) as approved by the Independent Ethics Committee (IEC), before any screening evaluations.
* Male subjects between 30 to 64 years of age (extremes included), on the date of signing the ICF.
* A body mass index between 18 to 32 kg/m2 (extremes included).
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and fasting clinical laboratory safety tests, and not having had any clinically significant illness in the 3 months before first investigational medicinal product (IMP) administration.
* Having a regular and (at least) daily defecation pattern.
* Able and willing to comply with restrictions on prior and concomitant medication as described in the protocol.
* Nonsmoker, defined as an individual who has abstained from smoking (or the use of e-cigarettes or nicotine containing products) from at least 2 months before screening. Having a breath carbon monoxide reading of ≤10 parts per million.
* Negative urine drug screen (e.g. amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, tricyclic antidepressants) and alcohol breath test.
* Male subjects with female partners of childbearing potential willing to comply with the contraceptive methods described in the protocol from the time of the first IMP administration, during the clinical study, and for at least 90 days after the last IMP administration.

Exclusion Criteria:

* Known hypersensitivity to IMP ingredients or history of a significant allergic reaction to IMP ingredients as determined by the investigator, such as anaphylaxis requiring hospitalization, and/or known sensitivity to IMP or the excipients (e.g. lactose). Hayfever is allowed unless active.
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) antibody, or history of hepatitis from any cause with the exception of a history of hepatitis A infection at least 12 weeks before first IMP administration.
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus [HIV] infection).
* Presence or sequelae of gastrointestinal, liver, kidney (creatinine clearance ≤80 mL/min, using the Cockcroft-Gault formula), or other conditions known to interfere with the absorption, distribution, metabolism, and excretion (ADME) properties of drugs. Subjects with documented Gilbert's syndrome are eligible for inclusion in the study.
* History of malignancy within the past 5 years (except for basal cell carcinoma of the skin that has been treated and with no evidence of recurrence).
* Hemoglobin level below the lower limit of normal (LLN; 13.0 g/dL). Retesting is allowed once.
* Significant blood loss (including blood donation [>450 mL]) or transfusion of any blood product within 12 weeks before screening.
* Active drug abuse (per investigator judgment) or alcohol abuse (more than three glasses of wine, beer, or equivalent/day) within 3 months before first IMP administration.
* Concurrent participation or participation in a drug, drug/device or biologic investigational research study within 12 weeks or 5 half-lives of the drug, whichever is longer, before first IMP administration.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic Xrays and other medical exposures, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, can participate in the study.

Ages: 30 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Change of total radioactivity excreted in urine and feces combined (µg) from baseline at Day 10 (Part 2) | From Day 1 pre-dose up to Day 10
  To assess the mass balance using [14C]-GLPG1690.
Maximum observed plasma concentration (Cmax) of total radioactivity (Part 2). | From Day 1 pre-dose up to Day 10
  To assess the pharmacokinetics (PK) of GLPG1690 and its main metabolites in plasma
Maximum observed plasma concentration (Cmax) of GLPG1690 (Part 2). | From Day 1 pre-dose up to Day 10
  To assess the pharmacokinetics (PK) of GLPG1690 and its main metabolites in plasma
Area under the plasma concentration-time curve (AUC) of total radioactivity (Part 2). | From Day 1 pre-dose up to Day 10
  To assess the PK of GLPG1690 and its main metabolites in plasma
Area under the plasma concentration-time curve (AUC) of GLPG1690 (Part 2). | From Day 1 pre-dose up to Day 10
  To assess the PK of GLPG1690 and its main metabolites in plasma
Change in amount of [14C] GLPG1690 excreted in urine and feces combined (µg) from baseline at Day 7 (Part 2). | From Day 1 pre-dose up to Day 7
  To better characterize the elimination pathways and metabolite profile of GLPG1690

SECONDARY OUTCOMES:
Intravenous (IV) maximum observed plasma concentration (Cmax) of [14C]-GLPG1690 microtracer (MT) (Part 1). | From Day 1 pre-dose up to Day 4
  To assess the PK of GLPG1690 and its main metabolites in plasma.
Intravenous (IV) maximum observed plasma concentration (Cmax) of total radioactivity (Part 1). | From Day 1 pre-dose up to Day 4
  To assess the PK of GLPG1690 and its main metabolites in plasma.
IV Area under the plasma concentration-time curve (AUC) of [14C]-GLPG1690 microtracer (MT) (Part 1). | From Day 1 pre-dose up to Day 4
  To assess the PK of GLPG1690 and its main metabolites in plasma.
IV Area under the plasma concentration-time curve (AUC) of total radioactivity(Part 1). | From Day 1 pre-dose up to Day 4
  To assess the PK of GLPG1690 and its main metabolites in plasma.
Safety and tolerability of GLPG1690, assessed by the number of subjects with adverse events (AEs) (Part 1 and Part 2). | From screening through study completion, an average of 2 months
  To evaluate the safety and tolerability of GLPG1690 (in Part 1 and Part 2).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brearley, BM. MRCP, Study Director — Galapagos NV
Locations (1):
- Quotient Sciences Limited, Ruddington, United Kingdom